CLINICAL TRIAL: NCT04004247
Title: Effects of High Flow Nasal Cannula on Breathing and the Respiratory System Parameters
Acronym: HaFo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HFNC-01
Record Dates: First submitted 2019-06-16; First posted 2019-07-02 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: High Flow Oxygenation; Electrical Impedance Tomography; Non invasive ventilation

STUDY DESIGN:
Intervention Model Description: 12 volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 10-12 young healthy volunteers. Placed on semi-sitting position on the bed (40 deg.elevation). Calibration of electrical impedance tomography (EIT) on defined tidal volume 500ml, done with 500ml syringe connected to closed breathing circuit using full face mask as an interface.
  Insertion an esophageal and nasopharyngeal catheter for pressures measurement. In the first phase - spontaneous breathing with full face mask at 0, 5 and 10 cm H20 levels of PEEP.
  In the second phase - high flow oxygenation through nasal cannula, start with flow rate 10 L/min with gradual increase up to 60 L/min.
  Spirometry to determine functional residual capacity (FRC) before and after procedure is planed.
  Interventions: Device: High Flow Nasal generator (AirVO2)

INTERVENTIONS:
Device: High Flow Nasal generator (AirVO2) — High Flow Nasal Oxygenation
  Other Names: Full face mask connected to ventilator (Avea)

SUMMARY:
The aim of this study is a detailed investigation of the effect of High Flow Nasal Oxygenation (HFNO) on respiratory system characteristics and ventilation parameters in healthy adult subjects and the subsequent use of measured data to answer the following questions:

What level of positive end expiratory pressure (PEEP) causes a HFNO with different flow rates? Does HFNO work as pressure support or does it act more like a Continuous Positive Airway Pressure (CPAP) ventilation?

DETAILED DESCRIPTION:
High Flow Oxygen through nasal cannula is widely used in the setting of hypoxemic respiratory failure of heterogenous etiology with very good patients compliance.

However, the evidence of what level of PEEP or pressure support (if any) with different flow rates is weak.

Our goal is to determine these effects and compare them with standard approach with non-invasive ventilation via full face mask.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers willing to participate

Exclusion Criteria:

* general contraindications for oesophageal catheter insertion: oesophageal varices, bleeding disorders (including anticoagulant medication), diverticulitis, oesophageal tumors, history of recent oesophageal/gastric surgery, recent epistaxis,
* sinusitis
* allergy to local anesthetics
* subject refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Measurement of inspiratory pressure, pressure in a hypopharynx and pleural pressure estimation using oesophageal catheter on conventional non-invasive ventilation (NIV). | 1 hour
  Using measurement of several pressures - inspiratory, oesophageal, nasopharyngeal (cm of H20 on conventional NIV.
Measurement of inspiratory pressure, pressure in a hypopharynx and pleural pressure estimation using oesophageal catheter on High flow nasal oxygenation (HFNO). | 1 hour
  Using measurement of several pressures - inspiratory, oesophageal, nasopharyngeal (cm of H20) on High flow nasal oxygenation (HFNO).
Calculation of Pressure Time Product (PTP) for estimation of Work of Breathing (WOB). | up to 8 weeks
  Compare PTP between conventional NIV and HFNO.
Monitoring of EIT during spontaneous ventilation on conventional non-invasive ventilation (NIV). | 1 hour
  EIT for description of distribution of ventilation on conventional NIV at different levels of PEEP (cm H20).
Monitoring of EIT during spontaneous ventilation with High flow nasal oxygenation (HFNO). | 1 hour
  EIT for description of distribution of ventilation with HFNO with different flow rate levels (litres per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Michal Sotak, MD., DESA, Principal Investigator — Military University Hospital, Prague; Jan Filip, Principal Investigator — Czech Technical University in Prague
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355